CLINICAL TRIAL: NCT05421897
Title: RAPID Feasibility Study: A Pilot Study for the Rapid Infusion of Dinutuximab
Brief Title: Rapid Administration Pilot for Infusing Dinutuximab
Acronym: RAPID
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Principal Investigator, Sara-Jane Onyeama, Assistant Professor, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-22-00205; NCI-2025-06180 (Other: NCI Trial Identifier)
Record Dates: First submitted 2022-06-08; First posted 2022-06-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-10

CONDITIONS: Neuroblastoma
Keywords: relapsed neuroblastoma; refractory neuroblastoma; persistent high-risk neuroblastoma; pediatric cancer
MeSH Terms: conditions — Neuroblastoma; Neoplasms | interventions — dinutuximab; Drug Therapy; Cyclophosphamide; Topotecan; Temozolomide; Irinotecan; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rapid infusion of dinutuximab with chemotherapy (Experimental): Patients will receive chemotherapy and dinutuximab via rapid infusion
  Interventions: Drug: Dinutuximab with Chemotherapy

INTERVENTIONS:
Drug: Dinutuximab with Chemotherapy — Rapid infusion of dinutuximab in 5 hours or less
  Other Names: Cyclophosphamide; Topotecan; Temozolomide; Irinotecan; Sagramostim

SUMMARY:
Studies have shown that the anti-GD2 human-mouse chimeric monoclonal antibody dinutuximab has contributed significantly to the improvement of treatment for children with high-risk neuroblastoma and has become a mainstay in treating high risk neuroblastoma in children as part of up-front therapy and relapsed/refractory therapy. The administration of dinutuximab requires a significant amount of time and resources to complete the 10-20 hour standard infusion time for 4 days in the inpatient setting. During its early development, a phase I study profiling the clinical efficacy and tolerability of dinutuximab infusions in children successfully infused dinutuximab at various rates including over 1 hour at different dose levels. In the adult setting, dinutuximab has been tolerated over substantially shorter infusion times (less than 2 hours). Additionally, another anti-GD2 murine monoclonal antibody naxitamab, which has a similar toxicity profile to dinutuximab, is FDA approved for administration over 90 minutes and is successfully administered in outpatient setting. Given this reassuring data the investigators aim to evaluate the feasibility of the rapid administration of dinutuximab over four hours or less in our patient population of children with high-risk neuroblastoma. The pharmacokinetics, toxicity profile and supportive care requirements will be analyzed and described in order to determine if rapid infusion of dinutuximab can be successfully tolerated over four hours or less which would allow for administration of this agent in the outpatient setting. Should this trial prove to be successful, it would serve to decrease the hospital burden in a positive way by allowing for administration of this immunotherapy agent in the outpatient setting and patients may prefer shorter infusion duration. Furthermore, it could lessen overall costs and inpatient admissions for patients.

DETAILED DESCRIPTION:
Neuroblastoma is the most common extracranial solid tumor of childhood. While it comprises only 8% of all childhood cancer cases, neuroblastoma is responsible for 12% of cancer deaths in children under 15 years of age. Approximately 50% of neuroblastoma patients are classified as high-risk, and over half of these children succumb to their disease despite intensive multi-modal therapy. The prognosis is worse for patients whose disease is refractory to initial therapy or who experience a recurrence of their tumor, as the majority of these patients cannot be cured of their disease. However, rates of event free survival and overall survival have improved over the past decades with the introduction of dinutuximab.

Dinutuximab is a chimeric monoclonal antibody that targets disialoganglioside (GD2) receptors. It has become an integral modality in the treatment of high-risk neuroblastoma (HR NBL) in up-front therapy and in the setting of relapsed or refractory disease. Additionally, there are numerous ongoing trials that include dinutuximab as part of the backbone therapy or in combination with other agents to improve tumor response in HR NBL patients.

A limiting factor for the use of dinutuximab has been the management of infusion-related toxicities. GD2 is expressed on neurons, skin melanocytes, and peripheral pain fibers of human tissues, which is evident in the common manifestation of pain during infusions. Other most common adverse effects include hypotension, capillary leak syndrome, and infusion-related reactions. These toxicities typically last during the standardized infusion duration of 10-20 hours but typically do not correlate with plasma levels. Pain that occurs during the infusion typically resolves shortly after the infusion is completed, despite the fact that dinutuximab persists in the circulation, which suggests that pain may be related to infusion rate rather than drug exposure (AUC). Due to the lengthy infusion duration and high frequency of side effects, dinutuximab infusions currently require significant hospital resources including nursing care, opioid infusions, around the clock supportive care medications, and a hospital stay for a minimum of 4-5 days.

With the expectation of repeated cycles of dinutuximab for different protocols in HR NBL treatment and with the expansion of dinutuximab studies in other GD2 positive tumors, there is a need to improve the administration and management of dinutuximab for future practicality and patient durability. A different anti-GD2 antibody naxitamab with a similar side effect profile to dinutuximab has been FDA approved for administration in the outpatient setting. Therefore, there is potential for dinutuximab to be administered in the outpatient setting. Although some studies have attempted to modify the administration of dinutuximab dosing and infusion durations, none have focused on shortening infusion time in the pediatric setting.

Dinutuximab was shown to significantly improve survival in children with HR NBL when administered after dose-intensive combination chemotherapy and high-dose myeloablative therapy with autologous stem cell rescue, and when combined with immunomodulating agents sargramostim and aldesleukin (IL-2) in the randomized phase 3 clinical trial, ANBL 0032. This Children's Oncology Group (COG) trial found that the combination of dinutuximab with sargramostim and IL-2 enhanced antibody-dependent cell-mediated cytotoxicity when given with isotretinoin in post-consolidation therapy. The addition of immunotherapy to isotretinoin in the post-consolidation phase was found to be significantly superior to isotretinoin alone. This led to the FDA approval of dinutuximab in the post-consolidation setting of neuroblastoma therapy. More recently, when dinutuximab was combined with irinotecan, temozolomide and sargramostim in patients with relapsed/refractory neuroblastoma (ANBL 1221) improved response rates were seen and as a result, this regimen is now considered first line for patients with relapsed or refractory disease in North America.

In 2019, the COG Neuroblastoma Committee released a memo removing IL-2 from the standard care for post-consolidation immunotherapy in HR NBL patients. The memo cited the data from two studies by the International Society of Pediatric Oncology Europe Neuroblastoma (SIOPEN) that showed no difference in survival outcomes with the inclusion of IL-2. This led to IL-2 elimination from both SIOPEN and COG protocols. Ongoing trials of post-consolidation immunotherapy were adopted to reflect this update but there are no completed clinical trials reporting data of dinutuximab with sargramostim without chemotherapy or IL-2.

The current dose of dinutuximab is 17.5mg/m2/day given over 10 hours for 4 days. It is typically given with pre-medications, opiates and supportive care with careful monitoring of AE's and early intervention as needed. The infusion rate may be slowed down but needs to be completed in 20 hours. Since the published results of dinutuximab efficacy in neuroblastoma and with many years of experience administering it, patients have been successfully completing many courses of therapy in the relapsed setting with good control of AE's.

Initially the A0935A protocol directed dinutuximab infusion over 10 hours but was then revised to be given over 5 hours based on tolerability. The ANBL 0032 protocol directed the infusion of dinutuximab over 6 hours. This was suspended temporarily in 2009 for an investigation into the apparent increase in allergy-like AEs related to IL-2; the protocol was amended to extend the dinutuximab infusion duration to 10-20 hours. However since IL-2 removal from standard protocols in 2019, no studies have evaluated the tolerability of infusing dinutuximab in under 10 hours in the HR NBL patient population.

Based on clinical experience of infusing this agent at Children's Hospital Los Angeles (CHLA), the peak time for capillary leak and worsening pain occurs at or after 4 hours of dinutuximab infusing. Therefore, it is reasonable to conclude that fast infusion may ameliorate some of the symptoms experienced by patients.

Although dinutuximab has most recently been given in 10-20 hour infusions based on the ANBL0032 study data that included IL-2, the experience of the early studies of dinutuximab with shorter infusion rates, and the fact that similar anti-GD2 antibodies such as Naxitamab and Hu14.18k322A, are well tolerated in 4 hours or less, support further investigation into decreasing the infusion time of dinutuximab in pediatric patients. The inclusion of this agent in the upfront and relapse settings of neuroblastoma therapy highlights the impact this pilot study would have. If successful in the pilot setting, this could be incorporated into larger-scale studies.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients ≥ 12 months of age at the time of enrollment are eligible for this study.
* Diagnosis: Patients must have a diagnosis of relapsed , refractory (defined as achieving less than a partial response), or persistent high risk neuroblastoma or ganglioneuroblastoma (nodular) [verified by tumor pathology analysis or demonstration of clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites at the time of diagnosis] and have been designated as having high-risk disease based on COG risk classification.

No minimal sites of disease are required for this study.

Prior Therapy (all timeframes below apply from time of enrollment):

* Must have completed high-risk Induction therapy with at least 4 cycles of chemotherapy.
* At least 14 days must have elapsed since completion of myelosuppressive therapy.
* Patients must have received previous treatment with dinutuximab (with or without chemotherapy).
* Anti-cancer agents not known to be myelosuppressive (e.g. not associated with substantially reduced platelet or ANC counts) are permitted while on study with PI approval. However, they must be held during protocol therapy. The anti-cancer agent may be resumed after completion of final dinutuximab day in each cycle per physician discretion.
* Antibodies: ≥ 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to Grade ≤ 1.
* Immnoglobulins: IVIG should not be given within 2 weeks of starting dinutuximab treatment and 1 week after completing dinutuximab therapy.
* Patients must have been off pharmacologic doses of systemic steroids for at least 7 days prior to enrollment.
* Patients who require or are likely to require pharmacologic doses of systemic corticosteroids while receiving treatment on this study are ineligible. (The only exception is for patients known to require 2mg/kg or less of hydrocortisone, or an equivalent dose of an alternative corticosteroid, as premedication for blood product administration in order to avoid allergic transfusion reactions). The use of conventional doses of inhaled steroids for the treatment of asthma is permitted, as is the use of physiologic doses of steroids for patients with known adrenal insufficiency.
* Radiation may be given up to 1 week prior to enrollment if clinically indicated. Palliative radiation while on study is permitted but not during infusion days.
* Stem cell transplant must be >6months prior to enrollment. Patients who received autologous stem cell infusion to support non-myeloablative therapy (such as 131 I-MIBG) are eligible at any time as long as they meet the other criteria for eligibility.
* 131I-MIBG therapy: Patients are eligible ≥6 weeks after therapeutic 131I-MIBG provided that all other eligibility criteria are met.
* Prior or planned concomitant treatment with eculizumab is permitted (e.g., treatment of TA-TMA).

Adequate Bone Marrow Function Defined As:

* Peripheral absolute neutrophil count (ANC) ≥750/microL
* Platelet count ≥50,000/mL (transfusion independent for prior 7 days). Exemptions may be granted for patient specific criteria (i.e. low platelet function due to history of extensive prior therapy or bone marrow disease)
* Hematologic growth factor may given up to 14 days prior to enrollment

Adequate Renal Function Defined As:

* Creatinine clearance or radioisotope GFR ≥70mL/min/1.73m2 or
* Adequate serum creatinine based on age/gender

Note: Patients with history of transplant-associated thrombotic microangiopathy (TA-TMA) must have a creatinine clearance or radioisotope GFR at baseline to assess renal function and must meet the above criteria.

Adequate Liver Function Defined As:

* Total bilirubin ≤1.5 x ULN for age AND
* SGPT (ALT) ≤ 5.0 x ULN for age (≤ 225 U/L). For the purpose of this study, the ULN for SGPT is 45U/L.

Adequate Central Nervous System Function Defined As:

* Patients with a history of CNS disease must have no clinical evidence of active progressive CNS disease at the time of study enrollment. Patients with history of CNS disease need to have at least stable tumor in the CNS for at least one month.
* Patients with seizure disorders may be enrolled if seizures are well controlled on antiepileptic medication
* CNS toxicity ≤ Grade 2

Adequate Cardiac Function Defined As:

* Shortening fraction of ≥27% by ECHO, or
* Ejection fraction of ≥50% by ECHO or gated radionuclide study.

Adequate Pulmonary Function Defined As: No evidence of dyspnea at rest, no exercise intolerance, no chronic oxygen requirement, and room air pulse oximetry >94% if there is a clinical indication for pulse oximetry. For patients who do not have respiratory symptoms, full PFTs are NOT required.

Exclusion Criteria:

* Men and women of childbearing potential and their partners must agree to use adequate contraception while enrolled on this study.
* Females of childbearing potential (≥ 10 years of age and /or post-menarchal) must have a negative pregnancy test to be eligible for this study, and they must agree to use 2 acceptable methods of contraception or abstain from heterosexual intercourse while participating in this study.
* Pregnant women will be excluded from this study.
* Female patients who are lactating must agree to stop breastfeeding or will otherwise be excluded from this study.
* Patients with uncontrolled hypertension are not eligible; uncontrolled hypertension is defined as sustained hypertension not well-controlled on blood pressure medication(s).
* If enrolling on Regimen A (temodar, irinotecan, dinutuximab arm only): patients must not have received enzyme-inducing anticonvulsants including phenytoin, phenobarbital, or carbamazepine for at least 7days prior to study enrollment. Patients receiving non-enzyme inducing anticonvulsants such as gabapentin, valproic acid, or levetiracetam will be eligible. Patients who have received drugs that are strong inducers or inhibitors of CYP3A4 within 7 days prior to study enrollment are not eligible. Patients must not have ≥ Grade 2 diarrhea
* Patients must not have been diagnosed with myelodysplastic syndrome or with any malignancy other than neuroblastoma.
* Patients must not have uncontrolled infection.
* Patients with a history of Grade 4 allergic reactions to anti-GD2 antibodies or reactions that required permanent discontinuation of the anti-GD2 therapy are not eligible.
* Patients who could not tolerate standard dose of dinutuximab infusion in 20 hour or less are not eligible.
* Patients with a significant intercurrent illness or disease of any major organ system that would impair their ability to withstand protocol therapy are not eligible

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Determine feasibility of administering dinutuximab in Cycle 1 | Day 1 of therapy until Day 21
  The number of dinutuximab days tolerated in 4 hours or less in Cycle 1 will be measured
Determine average dinutuximab infusion time in Cycle 1 | Day 1 of therapy until Day 21
  The infusion time of dinutuximab days administered on Days 1-4 will be measured and the average infusion time will be calculated for each dinutuximab day during Cycle 1.

SECONDARY OUTCOMES:
Determine feasibility of administering Dinutuximab in Cycle 2-6 in 4 hrs or less | Day 22 of study therapy until Day 126
  The number of dinutuximab days tolerated in 4 hours or less in Cycles 2-6 will be measured
Determine average dinutuximab infusion time in Cycles 2-6 | Day 22 of study therapy until Day 126
  The infusion time of dinutuximab days administered on Days 1-4 will be measured and the average infusion time will be calculated for each dinutuximab day during Cycle 2-6.

CONTACTS AND LOCATIONS:
Overall Officials: Sara-Jane Onyeama, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu AL, Gilman AL, Ozkaynak MF, London WB, Kreissman SG, Chen HX, Smith M, Anderson B, Villablanca JG, Matthay KK, Shimada H, Grupp SA, Seeger R, Reynolds CP, Buxton A, Reisfeld RA, Gillies SD, Cohn SL, Maris JM, Sondel PM; Children's Oncology Group. Anti-GD2 antibody with GM-CSF, interleukin-2, and isotretinoin for neuroblastoma. N Engl J Med. 2010 Sep 30;363(14):1324-34. doi: 10.1056/NEJMoa0911123. PMID 20879881
- [Background] Yu AL, Gilman AL, Ozkaynak MF, Naranjo A, Diccianni MB, Gan J, Hank JA, Batova A, London WB, Tenney SC, Smith M, Shulkin BL, Parisi M, Matthay KK, Cohn SL, Maris JM, Bagatell R, Park JR, Sondel PM. Long-Term Follow-up of a Phase III Study of ch14.18 (Dinutuximab) + Cytokine Immunotherapy in Children with High-Risk Neuroblastoma: COG Study ANBL0032. Clin Cancer Res. 2021 Apr 15;27(8):2179-2189. doi: 10.1158/1078-0432.CCR-20-3909. Epub 2021 Jan 27. PMID 33504555
- [Background] Mody R, Naranjo A, Van Ryn C, Yu AL, London WB, Shulkin BL, Parisi MT, Servaes SE, Diccianni MB, Sondel PM, Bender JG, Maris JM, Park JR, Bagatell R. Irinotecan-temozolomide with temsirolimus or dinutuximab in children with refractory or relapsed neuroblastoma (COG ANBL1221): an open-label, randomised, phase 2 trial. Lancet Oncol. 2017 Jul;18(7):946-957. doi: 10.1016/S1470-2045(17)30355-8. Epub 2017 May 23. PMID 28549783
- [Background] Desai AV, Fox E, Smith LM, Lim AP, Maris JM, Balis FM. Pharmacokinetics of the chimeric anti-GD2 antibody, ch14.18, in children with high-risk neuroblastoma. Cancer Chemother Pharmacol. 2014 Nov;74(5):1047-55. doi: 10.1007/s00280-014-2575-9. Epub 2014 Sep 12. PMID 25212536
- [Background] Marachelian A, Desai A, Balis F, Katzenstein H, Qayed M, Armstrong M, Neville KA, Cohn SL, Bush M, Gunawan R, Lim AP, Smith MA, Smith LM. Comparative pharmacokinetics, safety, and tolerability of two sources of ch14.18 in pediatric patients with high-risk neuroblastoma following myeloablative therapy. Cancer Chemother Pharmacol. 2016 Feb;77(2):405-12. doi: 10.1007/s00280-015-2955-9. Epub 2016 Jan 20. PMID 26791869
- [Background] Mody R, Yu AL, Naranjo A, Zhang FF, London WB, Shulkin BL, Parisi MT, Servaes SE, Diccianni MB, Hank JA, Felder M, Birstler J, Sondel PM, Asgharzadeh S, Glade-Bender J, Katzenstein H, Maris JM, Park JR, Bagatell R. Irinotecan, Temozolomide, and Dinutuximab With GM-CSF in Children With Refractory or Relapsed Neuroblastoma: A Report From the Children's Oncology Group. J Clin Oncol. 2020 Jul 1;38(19):2160-2169. doi: 10.1200/JCO.20.00203. Epub 2020 Apr 28. PMID 32343642